CLINICAL TRIAL: NCT05436977
Title: Synergy Between morpHOlogical and inflammatoRy Evaluation in Predicting Long-term Coronary Plaque Progression
Acronym: SHORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: University of Cambridge (Other); Centro per la Lotta Contro l'Infarto - Fondazione Onlus (Other)
Responsible Party: Principal Investigator, Nevio Taglieri, Principal Investigator, University of Bologna
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHORE_Bo_2020
Record Dates: First submitted 2022-06-01; First posted 2022-06-29 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-05

CONDITIONS: Acute Coronary Syndrome; Atherosclerosis; Inflammation; Coronary Artery Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Atherosclerosis; Inflammation; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The coronary OCT images acquired will be analyzed off-line by an independent imaging core laboratory (Euroimage Research, Rome, Italy), using validated review stations. OCT-defined plaque classification was performed according to an international consensus statement and validated criteria.
  PET-CT and CT coronary angiography images will be analyzed off-line in an experienced imaging laboratory by our collaborators at the University of Cambridge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: coronary OCT — Intermediate coronary lesions will be evaluated by OCT
Diagnostic Test: 68GaDOTATATE PET/CTCA — Intermediate coronary lesions will be evaluated by68GaDOTATATE PET/CTCA

SUMMARY:
Data from human autopsy studies have showed that thrombosis of a ruptured plaque with a large necrotic core, inflammatory cells and a thin fibrous cap, the so-called thin cap fibroatheroma (TCFA), represents the main mechanism for acute coronary syndrome (ACS). Optical coherence tomography (OCT) is an imaging technique that provides high-resolution, cross-sectional images of tissue in situ. The resolution of OCT (10 um) is appropriate for measuring a cap thickness less than65 μm, and even the plaque macrophage density. 68Ga-DOTA-(Tyr3)-octreotate/NaI3-octreotide(68Ga-DOTA-TATE/NOC) Positron Emission Tomography (PET)/Computed Tomography coronary angiography (CTCA), targeting the somatostatin receptor subtype-2 selectively expressed by M1 macrophages may show coronary inflammation. The SHORE protocol aims at evaluating the synergy between OCT and 68Ga-DOTA-TATE/NOC in predicting coronary plaque progression as assessed by CTCA

DETAILED DESCRIPTION:
ACS are the leading cause of mortality and morbidity in the western world. Despite recommended therapies, after experiencing an ACS episode patients still have an increased cardiovascular risk during follow up. In the CLIMA study OCT criteria of plaque vulnerability at non-culprit sites such as minimum luminal area <3.5mm2, fibrous cap thickness <75 µm, lipid arc extension >180° and macrophage infiltration was associated with an increased risk of cardiac death and myocardial infarction (HR 7.54, 95%CI 3.1-18.6).

Of the 36 OCT defined vulnerable plaques only 7 were associated with events showing a very low positive predictive value (19%). Yet, among the 577 plaques with macrophages accumulation only the 5.2% was associated with the endpoint. The lack of reliable information on plaque inflammation could represent the miss point to better link high risk plaques to plaque progression and/or rupture. Recent studies showed that inflammation in coronary plaques may be measured by means 68Ga-DOTATATE/PET targeting the somatostatin receptor subtype-2 selectively expressed by M1 macrophages.

Thus the investigators aim to evaluate the in vivo natural history of coronary plaques characterized from both the morphological (OCT) and inflammatory (68Ga-DOTATATE PET/CTCA) point of view in patients with ACS and at least 1 intermediated coronary lesion as assessed by FFR/iFR

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants > 50 years old
* Able to give written, informed consent and to lie flat
* Presentation of ACS within ~2 weeks
* At least 1 intermediate (30-80% diameter stenosis) non-culprit coronary artery lesion on angiography, managed medically as clinically indicated (i.e.: negative FFR/iFR)

Exclusion Criteria:

* Women of child bearing potential not using adequate contraception
* Contrast allergy or contrast-nephropathy
* Uncontrolled atrial fibrillation
* Chronic kidney disease (eGFR <30 l/min/1.73m2)
* Uncontrolled chronic inflammatory disorder
* History of recent malignancy deemed relevant to the study by the investigator
* Current use of systemic corticosteroids
* Previous coronary artery bypass grafting surgery (CABG) or percutaneous coronary intervention (PCI) before the index event
* Contraindication to coronary angiography
* Requires CABG or staged non-culprit artery PCI
* Coronary vessels that could not be adequately imaged
* Severe valvular heart disease
* Any medical condition, in the opinion of the investigator, that prevents the participant from lying flat during scanning, or from participating in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Coronary Plaque Progression | 2 years
  Comparison of baseline non culprit OCT imaging and baseline 68Ga-DOTANOC tissue-to-blood ratio in patients with significant plaque progression measured by CTCA (defined by changes in low attenuation plaque volume and total atheroma volume), versus those without

SECONDARY OUTCOMES:
Coronary Plaque Progression | 2 years
  Comparison of baseline non culprit OCT imaging and 12 weeks 68Ga-DOTANOC tissue-to-blood ratio in patients with significant plaque progression measured at 2 years follow up by CTCA (defined by change in low attenuation plaque volume and total atheroma volume), versus those without

OTHER OUTCOMES:
Relationship between OCT and PET findings | baseline
  Comparison of 68Ga-DOTANOC imaging to OCT assessed plaque morphology

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bologna IRCCS Policlinico di St. Orsola, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
This protocol has been designed in collaboration with researchers in the United Kingdom, with the intention of combining data from the SHORE study with the Residual Inflammation and Plaque Progression Long-term Evaluation (RIPPLE; NCT04073810) study that is jointly sponsored by the University of Cambridge and Cambridge University Hospitals NHS Trust, UK.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after the recruiting phase and till the end of the study
Access Criteria: Only investigators of the Ripple study will have access to the data

REFERENCES:
- [Result] Prati F, Romagnoli E, Gatto L, La Manna A, Burzotta F, Ozaki Y, Marco V, Boi A, Fineschi M, Fabbiocchi F, Taglieri N, Niccoli G, Trani C, Versaci F, Calligaris G, Ruscica G, Di Giorgio A, Vergallo R, Albertucci M, Biondi-Zoccai G, Tamburino C, Crea F, Alfonso F, Arbustini E. Relationship between coronary plaque morphology of the left anterior descending artery and 12 months clinical outcome: the CLIMA study. Eur Heart J. 2020 Jan 14;41(3):383-391. doi: 10.1093/eurheartj/ehz520. PMID 31504405
- [Result] Tarkin JM, Joshi FR, Evans NR, Chowdhury MM, Figg NL, Shah AV, Starks LT, Martin-Garrido A, Manavaki R, Yu E, Kuc RE, Grassi L, Kreuzhuber R, Kostadima MA, Frontini M, Kirkpatrick PJ, Coughlin PA, Gopalan D, Fryer TD, Buscombe JR, Groves AM, Ouwehand WH, Bennett MR, Warburton EA, Davenport AP, Rudd JH. Detection of Atherosclerotic Inflammation by 68Ga-DOTATATE PET Compared to [18F]FDG PET Imaging. J Am Coll Cardiol. 2017 Apr 11;69(14):1774-1791. doi: 10.1016/j.jacc.2017.01.060. PMID 28385306